CLINICAL TRIAL: NCT04689503
Title: Study on the Measurement of Retinal Blood Flow in Children Based on Oct Angiography and the Effect of Optical Defocus Application
Brief Title: Study on the Measurement of Retinal Blood Flow in Children
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, vice-president, Wenzhou Medical University
Other Study IDs: retinal blood flow in children
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2019-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to provide reference for clinical application, the normal values of retinal blood flow parameters in Chinese healthy children were measured by oct-angiography. Meanwhile, the repeatability and consistency of retinal blood flow parameters measured by oct-angiography in children were further analyzed, and the correlation of retinal blood flow parameters with eye axis, choroidal thickness, age and diopter was analyzed, so as to provide basis for clinical diagnosis of children's ophthalmopathy. Objective to study the effect of short-term optical defocusing on retinal blood flow parameters, and analyze the correlation between the changes of posterior segment parameters before and after short-term optical defocusing, so as to provide the basis for the possible compensation mechanism of posterior segment optical defocusing, and further understand the possible physiological mechanism of myopia.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be 6-18 years old, with parents' consent and be able to abide by the experimental rules;
2. uncorrected visual acuity or spectacle corrected visual acuity ≥ 1.0, and each eye can fix the target;
3. equivalent spherical lens range + 0.50D ~ - 6.00D, binocular spherical lens anisometropia ≤ 1D, anisometropia ≤ 1.5D;
4. frame glasses can be worn for patients with ametropia, and hard contact lenses can not be worn for at least 4 weeks, and anisometropia can not be worn for 2 weeks
5. intraocular pressure in the normal range (9mmhg-21mmhg)

Exclusion Criteria:

1. Patients with history of ocular trauma and surgery;
2. patients with ocular organic lesions or systemic diseases;
3. patients with dry eye;
4. patients in the treatment period using drugs (such as atropine eye drops);
5. patients with poor cooperation or unqualified image quality

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children volunteers with normal corrected visual acuity
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Blood flow density measurement | 2017.05.01-2019.11.11
  The vascular density was defined as the percentage of the area occupied by the vascular cavity after secondary reconstruction. The percentage of vascular lumen in macular area is automatically displayed based on the early treatment of diabetic retinopathy study (ETDRS) partition (i.e. macular area, paramacular area, temporal area, last time area, nasal area and inferior area), and the other partition method is based on the "Nine Palace" partition (i.e. central macular area, supratemporal area, superior area, Supranasal area, nasal area, infranasal area, inferior area, infratemporal area and temporal area)

SECONDARY OUTCOMES:
Macular avascular area measurement | 2017.05.01-2019.11.11
  The new non vascular area measurement option was used to automatically measure the FAZ area. The boundary of avascular zone is detected and defined by system software and quantified automatically. The reference range of shallow retinal foveal avascular zone,It was defined as within 60 LM from the inner limiting membrane. In the images of shallow and deep capillary layers, the foveal avascular zone is measured automatically by clicking the center of foveal avascular zone.

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China